CLINICAL TRIAL: NCT07149194
Title: Assessment of the Accuracy of CBC-Derived Markers Against CRP and ESR in Detecting Active Rheumatoid Arthritis in Upper Egypt"
Brief Title: Accuracy of CBC Derived Markers Against CRP and ESR in Detecting Active Rheumatoid Arthritis in Upper Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abeer Hamdi Fahmi Abd Elhamid, Assessment of accuracy of CBC derived markers against CRP and ESR in detecting active Rheumatoid arthritis in upper Egypt, Assiut University
Other Study IDs: CBC markers in RA activity
Record Dates: First submitted 2025-08-24; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Rheumatoid arthritis
  Interventions: Other: CBC derived markers
- inactive Rheumatoid arthriti

INTERVENTIONS:
Other: CBC derived markers — CBC derived markers against CRP and ESR in detecting active Rheumatoid arthritis
  Groups: Active Rheumatoid arthritis

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease that leads to persistent synovial inflammation, joint destruction, and disability, often with extra-articular manifestations like interstitial pneumonia. It predominantly affects middle-aged individuals, especially women. Early diagnosis and accurate disease activity assessment are crucial to prevent irreversible joint damage and systemic complications (4).

Clinical tools like the Disease Activity Score in 28 joints (DAS28) are commonly used to monitor RA, relying on inflammatory markers such as C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR). However, CRP and ESR can be influenced by factors unrelated to RA, such as infections or anemia, and may not always be available or cost-effective in resource-limited settings (1).

In recent years, complete blood count (CBC)-derived markers have emerged as affordable and accessible alternatives for assessing systemic inflammation. These include the neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), lymphocyte-to-monocyte ratio (LMR), and red cell distribution width (RDW). These indices have shown strong correlations with RA disease activity in various studies, particularly NLR and RDW, which have high sensitivity and specificity for detecting active disease (2-3).

Studies in Egypt have explored the diagnostic accuracy of CBC-derived markers and composite indices like the CRP-to-albumin ratio (CAR) and albumin-to-fibrinogen ratio (AFR). These markers correlate significantly with DAS28 scores, suggesting they may be reliable indicators of RA disease activity in Egyptian patients (1-3).

ELIGIBILITY:
Inclusion Criteria:

* 1-Adults aged ≥18 years. 2-Established RA diagnosis according to ACR/EULAR criteria {ACR: American College of Rheumatology, a professional organization of rheumatologists.

EULAR: European League Against Rheumatism, a European organization for rheumatology.

3-Willing to provide informed consent

Exclusion Criteria:

* 1-Presence of infection, malignancy, or other autoimmune diseases. 2-Recent use (within 4 weeks) of corticosteroids or immunosuppressive therapy. 3-Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
the diagnostic accuracy of CBC-derived inflammatory markers in detecting active rheumatoid arthritis in Upper Egypt. | baseline
  the accuracy of CBC-derived inflammatory markers in diagnosis of active rheumatoid arthritis